CLINICAL TRIAL: NCT00318422
Title: Liraglutide Effect and Action in Diabetes (LEAD-1): Effect on Glycaemic Control After Once Daily Administration of Liraglutide in Combination With Glimepiride Versus Glimepiride Monotherapy Versus Glimepiride and Rosiglitazone Combination Therapy in Subjects With Type 2 Diabetes.
Brief Title: Effect of Liraglutide on Blood Glucose Control in Subjects With Type 2 Diabetes
Acronym: LEAD-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1436; 2005-003414-15 (EudraCT Number)
Record Dates: First submitted 2006-04-25; First posted 2006-04-26 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Rosiglitazone; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: liraglutide
Drug: rosiglitazone
Drug: glimepiride

SUMMARY:
This trial is conducted globally (the United States of America excepted). This trial is designed to show the effect of treatment with liraglutide when added to existing glimepiride therapy and to compare this to both glimepiride monotherapy and to rosiglitazone as add-on therapy to glimepiride.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Treatment with oral anti-diabetic drugs for at least 3 months
* HbA1c: 7.0-11.0 % (both incl.) in subjects on OAD monotherapy. 7.0-10.0 % (both incl.) in subjects on OAD combination therapy
* Body Mass Index (BMI) less than or equal to 45.0 kg/m2.

Exclusion Criteria:

* Treatment with insulin within the last three months
* Treatment with any drug that could interfere with the glucose level
* Any serious medical condition
* Females who are pregnant, have the intention of becoming pregnant or are breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1041 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 26 weeks of treatment

SECONDARY OUTCOMES:
body weight
Safety and tolerability
beta-cell function
Glycemic control parameters (fasting plasma glucose, -glucose profiles)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (107):
- Argentina (4):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Mar del Plata
  - Novo Nordisk Investigational Site, Mendoza
- Australia (9):
  - Novo Nordisk Investigational Site, Woolloongabba, Queensland
  - Novo Nordisk Investigational Site, Melbourne, Victoria
  - Novo Nordisk Investigational Site, Caboolture
  - Novo Nordisk Investigational Site, Ingleburn
  - Novo Nordisk Investigational Site, Kippa-Ring
  - Novo Nordisk Investigational Site, Miranda
  - Novo Nordisk Investigational Site, Randwick
  - Novo Nordisk Investigational Site, Southport
  - Novo Nordisk Investigational Site, Stones Corner
- Brazil (2):
  - Novo Nordisk Investigational Site, Fortaleza
  - Novo Nordisk Investigational Site, São Paulo
- Bulgaria (5):
  - Novo Nordisk Investigational Site, Pleven
  - Novo Nordisk Investigational Site, Plovdiv
  - Novo Nordisk Investigational Site, Rousse
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Varna
- Croatia (3):
  - Novo Nordisk Investigational Site, Osijek
  - Novo Nordisk Investigational Site, Slavonski Brod
  - Novo Nordisk Investigational Site, Split
- Czechia (5):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Ostrava
  - Novo Nordisk Investigational Site, Plzen - Lochotin
  - Novo Nordisk Investigational Site, Prague
- Finland (9):
  - Novo Nordisk Investigational Site, Espoo
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Lahti
  - Novo Nordisk Investigational Site, Nurmijärvi
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Pieksämäki
  - Novo Nordisk Investigational Site, Rauma
  - Novo Nordisk Investigational Site, Rovaniemi
  - Novo Nordisk Investigational Site, Tampere
- France (9):
  - Novo Nordisk Investigational Site, Dax
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Mougins
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Rennes
  - Novo Nordisk Investigational Site, Saint-Mandé
- Novo Nordisk Investigational Site, Athens, Greece
- India (4):
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Chandigarh, Punjab
  - Novo Nordisk Investigational Site, Chennai
  - Novo Nordisk Investigational Site, Mumbai
- Israel (3):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Italy (8):
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Lucca
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Napoli
  - Novo Nordisk Investigational Site, Perugia
  - Novo Nordisk Investigational Site, Ravenna
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Torino
- Malaysia (3):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Pulau Pinang
- Philippines (4):
  - Novo Nordisk Investigational Site, Davao City
  - Novo Nordisk Investigational Site, Makati City
  - Novo Nordisk Investigational Site, Marikina City
  - Novo Nordisk Investigational Site, Quezon City
- Poland (14):
  - Novo Nordisk Investigational Site, Bytom
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Gniewkowo
  - Novo Nordisk Investigational Site, Kamieniec Ząbkowicki
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Mazowieckie
  - Novo Nordisk Investigational Site, Nysa
  - Novo Nordisk Investigational Site, Rawa Mazowiecka
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Tychy
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Zabrze
- Romania (5):
  - Novo Nordisk Investigational Site, Brasov, Brașov County
  - Novo Nordisk Investigational Site, Ploieşti, Prahova
  - Novo Nordisk Investigational Site, Baia Mare
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Timișoara
- South Africa (3):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Umhlanga
- Novo Nordisk Investigational Site, Seoul, South Korea
- Spain (3):
  - Novo Nordisk Investigational Site, Gijón
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Reus
- Switzerland (4):
  - Novo Nordisk Investigational Site, Bern
  - Novo Nordisk Investigational Site, Lausanne
  - Novo Nordisk Investigational Site, Sankt Gallen
  - Novo Nordisk Investigational Site, Zurich
- Taiwan (3):
  - Novo Nordisk Investigational Site, Changhua
  - Novo Nordisk Investigational Site, Kaohsiung City
  - Novo Nordisk Investigational Site, Taipei
- Novo Nordisk Investigational Site, Bangkok, Thailand
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir

REFERENCES:
- [Result] Sullivan SD, Alfonso-Cristancho R, Conner C, Hammer M, Blonde L. Long-term outcomes in patients with type 2 diabetes receiving glimepiride combined with liraglutide or rosiglitazone. Cardiovasc Diabetol. 2009 Feb 26;8:12. doi: 10.1186/1475-2840-8-12. PMID 19245711
- [Result] Marre M, Shaw J, Brandle M, Bebakar WM, Kamaruddin NA, Strand J, Zdravkovic M, Le Thi TD, Colagiuri S; LEAD-1 SU study group. Liraglutide, a once-daily human GLP-1 analogue, added to a sulphonylurea over 26 weeks produces greater improvements in glycaemic and weight control compared with adding rosiglitazone or placebo in subjects with Type 2 diabetes (LEAD-1 SU). Diabet Med. 2009 Mar;26(3):268-78. doi: 10.1111/j.1464-5491.2009.02666.x. PMID 19317822
- [Result] Nauck M, Marre M. Adding liraglutide to oral antidiabetic drug monotherapy: efficacy and weight benefits. Postgrad Med. 2009 May;121(3):5-15. doi: 10.3810/pgm.2009.05.1997. PMID 19491535
- [Result] McGill JB. Insights from the Liraglutide Clinical Development Program--the Liraglutide Effect and Action in Diabetes (LEAD) studies. Postgrad Med. 2009 May;121(3):16-25. doi: 10.3810/pgm.2009.05.1998. PMID 19491536
- [Result] Blonde L, Russell-Jones D. The safety and efficacy of liraglutide with or without oral antidiabetic drug therapy in type 2 diabetes: an overview of the LEAD 1-5 studies. Diabetes Obes Metab. 2009 Dec;11 Suppl 3:26-34. doi: 10.1111/j.1463-1326.2009.01075.x. PMID 19878259
- [Result] Buse JB, Garber A, Rosenstock J, Schmidt WE, Brett JH, Videbaek N, Holst J, Nauck M. Liraglutide treatment is associated with a low frequency and magnitude of antibody formation with no apparent impact on glycemic response or increased frequency of adverse events: results from the Liraglutide Effect and Action in Diabetes (LEAD) trials. J Clin Endocrinol Metab. 2011 Jun;96(6):1695-702. doi: 10.1210/jc.2010-2822. Epub 2011 Mar 30. PMID 21450987
- [Result] Bode BW, Brett J, Falahati A, Pratley RE. Comparison of the efficacy and tolerability profile of liraglutide, a once-daily human GLP-1 analog, in patients with type 2 diabetes >/=65 and <65 years of age: a pooled analysis from phase III studies. Am J Geriatr Pharmacother. 2011 Dec;9(6):423-33. doi: 10.1016/j.amjopharm.2011.09.007. Epub 2011 Nov 4. PMID 22055210
- [Result] Henry RR, Buse JB, Sesti G, Davies MJ, Jensen KH, Brett J, Pratley RE. Efficacy of antihyperglycemic therapies and the influence of baseline hemoglobin A(1C): a meta-analysis of the liraglutide development program. Endocr Pract. 2011 Nov-Dec;17(6):906-13. doi: 10.4158/ep.17.6.906. PMID 22193143
- [Result] Hegedus L, Moses AC, Zdravkovic M, Le Thi T, Daniels GH. GLP-1 and calcitonin concentration in humans: lack of evidence of calcitonin release from sequential screening in over 5000 subjects with type 2 diabetes or nondiabetic obese subjects treated with the human GLP-1 analog, liraglutide. J Clin Endocrinol Metab. 2011 Mar;96(3):853-60. doi: 10.1210/jc.2010-2318. Epub 2011 Jan 5. PMID 21209033
- [Result] Zinman B, Schmidt WE, Moses A, Lund N, Gough S. Achieving a clinically relevant composite outcome of an HbA1c of <7% without weight gain or hypoglycaemia in type 2 diabetes: a meta-analysis of the liraglutide clinical trial programme. Diabetes Obes Metab. 2012 Jan;14(1):77-82. doi: 10.1111/j.1463-1326.2011.01493.x. Epub 2011 Oct 30. PMID 21883806
- [Result] Niswender K, Pi-Sunyer X, Buse J, Jensen KH, Toft AD, Russell-Jones D, Zinman B. Weight change with liraglutide and comparator therapies: an analysis of seven phase 3 trials from the liraglutide diabetes development programme. Diabetes Obes Metab. 2013 Jan;15(1):42-54. doi: 10.1111/j.1463-1326.2012.01673.x. Epub 2012 Sep 9. PMID 22862847
- [Result] Alves C, Batel-Marques F, Macedo AF. A meta-analysis of serious adverse events reported with exenatide and liraglutide: acute pancreatitis and cancer. Diabetes Res Clin Pract. 2012 Nov;98(2):271-84. doi: 10.1016/j.diabres.2012.09.008. Epub 2012 Sep 23. PMID 23010561
- [Result] King AB, Montanya E, Pratley RE, Blonde L, Svendsen CB, Donsmark M, Sesti G. Liraglutide achieves A1C targets more often than sitagliptin or exenatide when added to metformin in patients with type 2 diabetes and a baseline A1C <8.0%. Endocr Pract. 2013 Jan-Feb;19(1):64-72. doi: 10.4158/EP12232.OR. PMID 23186975
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- [Derived] Fonseca VA, Devries JH, Henry RR, Donsmark M, Thomsen HF, Plutzky J. Reductions in systolic blood pressure with liraglutide in patients with type 2 diabetes: insights from a patient-level pooled analysis of six randomized clinical trials. J Diabetes Complications. 2014 May-Jun;28(3):399-405. doi: 10.1016/j.jdiacomp.2014.01.009. Epub 2014 Jan 21. PMID 24561125
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com